CLINICAL TRIAL: NCT04406402
Title: The Effects of Different Acute Nutritional Protocols and Lifestyle Modification on Circulating L-arginine and Asymmetric Dimethylarginine (ADMA) in Obese and Type 2 Diabetic Subjects
Brief Title: L-arginine and Asymmetric Dimethylarginine (ADMA) and Lifestyle Protocols
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Wolfson Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 03
Record Dates: First submitted 2020-05-25; First posted 2020-05-28 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Diabetes Mellitus, Type 2; Obesity; Arginine; Asymmetric Dimethylarginine
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Acute glucose tolerance test (Experimental): A standard oral glucose tolerance test (75 grams of dextrose in 180 cc of water)
  Interventions: Behavioral: Acute dietary protocols and lifestyle modification
- Acute protein load test (Experimental): A protein-rich, vanilla-flavored powder (Pro-gym, Telpharma, Is
  Interventions: Behavioral: Acute dietary protocols and lifestyle modification
- Acute fat load test (Experimental): a 100-gram portion of sweet cream containing 300 Kacls, of which 94% of the ingested calories were fat
  Interventions: Behavioral: Acute dietary protocols and lifestyle modification
- Acute alcohol load test (Experimental): Vodka (100 cc, 40% alcohol)
  Interventions: Behavioral: Acute dietary protocols and lifestyle modification
- Acute exercise (Experimental): 30 minutes of supervised graded walking on a treadmill according to each subject's individual ability. A goal heart rate was calculated as 70% of the age-adjusted maximal allowable heart rate.
  Interventions: Behavioral: Acute dietary protocols and lifestyle modification
- Lifestyle modification program - 12 weeks (Experimental): 12 weeks of weight-loss dietary program constructed according to the guidelines of the American Diabetes Association. Based on weight, gender, and age, daily dietary allowance varied at 1200-1800 Kcal, 50% carbohydrates, 20% protein, and 30% fat. Participants were also asked to engage in moderate physical activity comprised of a 40-minute walk three times a week. A weekly clinic visit alternating with a weekly telephone contact was also required.
  Interventions: Behavioral: Acute dietary protocols and lifestyle modification

INTERVENTIONS:
Behavioral: Acute dietary protocols and lifestyle modification — The investigators tested the effects on serum Arg and ADMA of a) a single load of ingested dextrose, protein, fat or alcohol, each consumed within 10 minutes; b) a single episode of physical exercise; c) a 12 weeks lifestyle modification program comprised of a standard dietary and physical activity counseling in obese or T2DM subjects on circulating Arg and ADMA (n=43).

SUMMARY:
Low serum L-arginine (Arg) and high asymmetric dimethylarginine (ADMA) can predict microvascular complications in type 2 diabetes (T2DM). The investigators examined whether or not Arg and ADMA are affected by dietary factors or lifestyle modification in overweight/ obese and T2DM subjects.

DETAILED DESCRIPTION:
The investigators tested the effects on serum Arg and ADMA of a) a single load of ingested dextrose, protein, fat or alcohol, each consumed within 10 minutes; b) a single episode of physical exercise; c) a 12 weeks lifestyle modification program comprised of a standard dietary and physical activity counseling in obese or T2DM subjects on circulating Arg and ADMA (n=43)

ELIGIBILITY:
Inclusion Criteria:

* obese and/ or T2DM subjects

Exclusion Criteria:

* type 1 diabetes
* insulin-treated T2DM
* active coronary disease (recent [≤ 6months] myocardial infarction, unstable angina, recent coronary catheterization, or coronary bypass grafting
* individuals with significant impairment in liver enzymes (≥ 2.5 the upper limit of the normal range)
* serum creatinine higher than 1.5mg%
* known malabsorption, alcoholism or illicit use of drugs
* abnormal thyroid function tests
* concomitant or recent use of glucocorticoids
* uncertain mental state (to avoid invalid informed consent or lack of compliance).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2006-12-05 (Actual); Primary Completion 2008-04-04 (Actual); Study Completion 2008-12-10 (Actual)

PRIMARY OUTCOMES:
Serum L-arginine change | For acute phase: before the nutritional/exercise load (time 0), as well as 30, 60, 90, 120 and 150 minutes after the challenge test. And from baseline to 12 weeks for lifestyle modification phase
  Change in arginine levels (absolute and relative) (µmol/l)
High asymmetric dimethylarginine (ADMA) change | For acute phase: before the nutritional/exercise load (time 0), as well as 30, 60, 90, 120 and 150 minutes after the challenge test. And from baseline to 12 weeks for lifestyle modification phase
  Change in ADMA levels (absolute and relative) (µmol/l)

SECONDARY OUTCOMES:
Body mass index (BMI) change | From baseline to 12 weeks for lifestyle modification phase
  Change in BMI levels (Kg/m2)
Glycated hemoglobin (HbA1c) change | From baseline to 12 weeks for lifestyle modification phase
  Change in HbA1c levels (%)

CONTACTS AND LOCATIONS:
Overall Officials: Naftali Stern, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Diabetes Unit, E. Wolfson Medical Center, Holon, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buch A, Ganz T, Wainstein J, Gilad S, Limor R, Shefer G, Boaz M, Stern N. Alcohol Drinks Induce Acute Lowering in Circulating l-Arginine in Obese and Type 2 Diabetic Subjects. J Med Food. 2022 Jun;25(6):675-682. doi: 10.1089/jmf.2021.0045. PMID 35708634